CLINICAL TRIAL: NCT04808453
Title: A Phase 1, First-in-Human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of CPI-300 Via Intravenous Infusion in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of CPI-300 in Patients With Advanced Tumors
Acronym: CPI-300
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coordination Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPI-300CL21-01
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Advanced Tumors
Keywords: Intravenous Infusion

STUDY DESIGN:
Intervention Model Description: accelerated titration method followed by a conventional 3 + 3 dose escalation study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPI-300 (Experimental): Dose Escalation Group: CPI-300 will be administered via intravenous infusion once every 2 weeks for up to 6 dose levels using an accelerated titration method followed by a conventional 3 + 3 study design
  Interventions: Drug: CPI-300

INTERVENTIONS:
Drug: CPI-300 — CPI-300 will be administered via intravenous infusion on Day 1 of a 14-Day cycle

SUMMARY:
This is a prospective, open-label, single arm, non-randomized study of CPI-300 in patients with advanced tumors. CPI-300 is administered via intravenous infusion using an accelerated titration method followed by a conventional 3 + 3 study design to identify the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
Up to 6 dose levels of CPI-300 will be tested. MTD will be defined as the dose associated with a dose limiting toxicity (DLT) in less than or equal to 33% of patients at the dose level tested. Dose limiting toxicity (DLT) is defined as one of the following events occurring from the intravenous injection of CPI-300 within 28 days:

* Grade 4 or greater treatment related adverse events
* Any Grade 3 or greater treatment related non-hematologic, non-dermatologic toxicity (including nausea, vomiting or diarrhea lasting more than 72 hours)

Blood samples will be drawn to determine drug blood concentrations for pharmacokinetic assessment.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically confirmed diagnosis of advanced solid tumor
* Have advanced or metastatic disease refractory to standard curative or palliative therapy or contraindication to standard therapy
* Have an ECOG performance status of 0-1
* Have adequate bone marrow reserve, liver and renal function
* Be reasonably recovered from preceding major surgery or no major surgery within 4 weeks prior to the start of Day 1 treatment
* Have a negative pregnancy test for females with child bearing age at screening and should not be breast feeding
* Be willing to abstain from sexual activity or practice physical barrier contraception from study entry to 6 months after the last day of treatment

Exclusion Criteria:

* Have peripheral neuropathy of Grade 3 or Grade 4 at screening
* Have peripheral sensory neuropathy of Grade 2 or greater at screening
* Have an interval from previous neurotoxic drugs less than 3 months unless reasonably recovered from all grades of neurotoxicity to grade 1 or lower as judged by the investigator
* Have known hypersensitivity to chemotherapeutic agents
* Have chronic diarrhea
* Have a history of thrombocytopenia with complications including hemorrhage or bleeding > Grade 2 that required medical intervention or any hemolytic condition or coagulation disorders that would make participation unsafe
* Have unresolved toxicity from previous treatment or previous investigational agents; excluding alopecia
* Received investigational agents or systemic anticancer agents (other than neurotoxic compounds) within 5 half lives or 28 days, whichever is shorter, prior to Day 1 of treatment
* Have signs or symptoms of end organ failure, major chronic illnesses other than cancer, or any severe concomitant conditions
* Have experienced any of the following within the 6-month period prior to screening: angina pectoris, coronary artery disease or cerebrovascular accident, transient ischemic attack, cardiac failure with known ejection fraction less than 40%, or cardiac arrhythmia requiring medical therapy
* Have other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that would make the patient inappropriate for enrollment in this study
* Is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 28 days
  To determine the maximum tolerated dose (MTD), which is defined as the highest dose level at which number of patients reporting a dose limiting toxicity (DLT) is less than or equal to 33%

SECONDARY OUTCOMES:
Clinical Benefit | 28 Days and additional CPI-300 treatments till disease progression or intolerability
  To assess clinical benefit by response rate and resolution of symptoms, which will be reported as response rate (%)
Adverse Effect | 28 Days and additional CPI-300 treatment till disease progression or intolerability
  To assess adverse effect as either treatment-related or non-treatment-related as defined by CTCAE
Maximum Plasma Concentration (Cmax) | 8 Days
  To evaluate maximum plasma concentration (Cmax) of CPI-300 in patients tested
Area Under the Curve (AUC) | 8 Days
  To evaluate area under the curve (AUC) of CPI-300 in patients tested

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Florida Cancer Specialists, Lake Mary, Florida
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No